CLINICAL TRIAL: NCT05993117
Title: Rechargeable Implantable Vagus Nerve Stimulation System for Drug-Refractory Epilepsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Pins Medical Co., Ltd (Industry)
Collaborators: Peking University First Hospital (Other); Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PINS-VNS-2101
Record Dates: First submitted 2023-07-28; First posted 2023-08-15 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Drug-Refractory Epilepsy
Keywords: Vagus Nerve Stimulation
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- G114R VNS system (Experimental)
  Interventions: Device: G114R VNS system

INTERVENTIONS:
Device: G114R VNS system — All patients treated with Rechargeable Implantable Vagus Nerve Stimulation System (G114R)

SUMMARY:
To evaluate the performance of automatic stimulation mode of a new rechargeable implantable vagus nerve stimulation system for drug-refractory epilepsy

DETAILED DESCRIPTION:
The study is a prospective, single-group, open-lable trial designed to collect data on patients implanted with a Model G114R VNS system (Beijing PINS Medical) from baseline through an EMU (epilepsy monitoring unit) stay of up to 5 days, and 3-mouth follow-up. The seizure burden and quality of life were evaluated. Adverse events were recorded during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥3 years old; gender is not limited;
* Patients with clinically diagnosed drug-resistant epilepsy, suitable for vagus nerve stimulation therapy;
* At least 6 seizures per month;
* Patients with a history of increased heart rate (tachycardia) associated with seizure onset based on clinical data obtained from medical history, admission/hospital charts, or prior neurophysiologic evaluations;
* When the patient is lying on the left side and in an upright position, from the proposed electrode position on the neck to the proposed pulse generator on the chest, the peak-peak R-wave of the ECG should be higher than 0.40mV;
* Patients who are willing to undergo EMU phase assessment and activate the automatic mode function during this period;
* Patients must be in good general health and ambulatory;
* Children and guardians must be willing and able to give informed consent;
* Patients and their families have good compliance and can cooperate with the completion of postoperative follow-up requirements.

Exclusion Criteria:

* Patients have had a bilateral or left cervical vagotomy;
* One or both sides of the vagus nerve have lesions or damage;
* Patients have a history of VNS Therapy;
* Patients with a history of status epilepticus within 1 year prior to enrollment;
* Patients with a history of mental illness or pseudoepileptic seizures or epilepsy caused by intracranial space-occupying lesions;
* Patients currently use, or are expected to use, short-wave diathermy, microwave diathermy, or therapeutic ultrasound diathermy;
* Patients expected to require full body magnetic resonance imaging;
* VNS therapeutic system implants will bring unacceptable surgical or medical risks to patients (according to the judgment of the investigator);
* Patients with surgical contraindications identified by surgeons and anesthesiologists such as tumors, insulin-dependent diabetes mellitus or poor general condition;
* A record of clinically significant seizure-related bradycardia (heart rate below 50 bpm);
* Patients prescribed drugs specifically for a cardiac or autonomic disorder that in the investigator's opinion would affect heart rate response unless the patient has ictal tachycardia while taking said drugs. These include, but are not limited to, beta adrenergic antagonists ("beta blockers");
* Patients with known clinically significant arrhythmias, and patients with clinically significant arrhythmias identified by 24-hour ambulatory ECG recordings obtained at the screening visit;
* Adult patients with severe mental illness, severe cognitive impairment, history of severe depression, or suicidal tendencies, which, in the judgment of the investigator, would pose an unacceptable risk to the patient or prevent the patient from successfully completing the study;
* Abusing alcohol or use narcotic drugs;
* Women who are pregnant. Women of childbearing age must take a pregnancy test;
* Patients currently enrolled in another investigational study;
* Those deemed unsuitable by the researcher.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of epilepsy detection | 2-4 weeks after implant
  Sensitivity is defined as the total number of seizures detected divided by the total number of seizures during the EMU stay.
False positives for epilepsy detection | 2-4 weeks after implant
  A false positive event is defined when the IPG judged a seizure and triggered automatic mode stimulation ±2 minutes outside the time window of a actual seizure. The ratio of the total number of false positive events for all subjects to the monitoring time for all subjects during the EMU phase is defined as the false positive rate.

SECONDARY OUTCOMES:
Changes in Seizure Frequency from Baseline | up to 3 months Visit
  Seizure frequency is calculated at 2 and 3 month follow-up visits based on seizure diary information and compared to baseline estimates. Response rate is computed and summarized for seizure as the percentage of patients that achieved ≥50% seizure reduction per month from baseline by visit.
Change in seizure Severity | up to 3 months Visit
  The Epilepsy Severity Scale (NHS3) will be completed at baseline，at the end of the EMU phase and during the follow-up period. The severity of epilepsy will be assessed based on seizure type. The range of NHS3 scale is 1-27 with 1 being the least severe and 27 being the most severe.
Change in Quality of Life | up to 3 months Visit
  Quality of life data is collected using patient-completed QOLIE-31 scales and compared between baseline and follow-up visits. The range for QOLIE-31-P (all subscores) is 0-100 with higher scores reflecting greater well-being.
Heart rate recording accuracy | 1 to 2 weeks after implantation
  The total number and accuracy of heart rate detected by IPG are measured by ECG recording.
Duty cycle | up to 3 months Visit
  The total percentage of time VNS is on for an individual patient is called the duty cycle. It's calculated as (ON time + X )/(ON time + OFF time), X depended on the setting of Soft start/stop.
Charging Equipment Satisfaction Evaluation | 2-4 weeks after implant
  A questionnaire is used to evaluate the simplicity of the charging process and overall satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Ye Wu, Principal Investigator — Peking University First Hospital; Jianguo Zhang, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China